CLINICAL TRIAL: NCT04119518
Title: Night Ambulatory Monitoring Of Blood Pressure Clinical Study Protocol
Brief Title: Night Ambulatory Monitoring Of Blood Pressure
Acronym: NAMBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-00614
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Intervention Model Description: Prospective, method-comparison, proof of concept, single centre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy and hypertensive subjects (Other): Subjects will be enrolled to be monitored for 24 hours via: the non-occlusive CSEM Pulse Watch, and a gold standard oscillometric device (Spacelabs OnTrak Ambulatory Blood Pressure monitor, Spacelabs Healthcare, Washington, USA) internationally validated for the 24h ABPM.
  Interventions: Device: CSEM Pulse Watch

INTERVENTIONS:
Device: CSEM Pulse Watch — Comparison of CSEM Pulse Watch with a gold standard oscillometric device Spacelabs OnTrak Ambulatory Blood Pressure monitor.

SUMMARY:
To determine accuracy of nightly non occlusive blood pressure measurements by the non-occlusive CSEM Pulse Watch compared to a gold standard oscillometric device Spacelabs OnTrak Ambulatory Blood Pressure monitor, Spacelabs Healthcare, Washington, USA) internationally validated for the 24h ABPM in Patients.

DETAILED DESCRIPTION:
Elevated Blood Pressure (BP) is a chronic medical condition with a prevalence of about 45% in the middle-aged population.

The particular interest of this project is given to the diagnosis and treatment of so-called nocturnal hypertension. Unfortunately, current monitoring practice relies on the use of occlusive pneumatic cuffs inflated around the arm to assess BP. Based on oscillometric technique, occlusive cuffs perform intermittent BP measurements every 20 minutes, thus providing only a limited view of the BP regulation landscape. In addition, oscillometric measurement performs a full occlusion of the measured arm inducing awakening reactions, and leading to non-representative overestimated BP values. The non-occlusive measurement of BP is thus an unsolved problem of modern medicine.

The aim of the NAMBP (Night Ambulatory Monitoring of Blood Pressure) project is to develop, implement and test in clinical trials a first-ever non-occlusive BP sensor to be used during sleep.

A novel technology for the non-occlusive measurement of BP from photoplethysmographic (optical) signals, known as Pulse Wave Analysis (PWA), has been investigated for the past decade by the Centre Suisse d'Electronique et de Microtechnique (CSEM, Neuchâtel, Switzerland). The herein proposed system - the CSEM Pulse Watch - consists in a single sensor (watch-like device) attached at the wrist that measures photoplethysmographic waveforms induced by the pulsatility of the skin arteries of the wrist. These waveforms are then post-processed via PWA: The system will detect features in the measured waveforms that correlate, through the phenomenon of wave reflections, to the underlying BP of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18y
* Good understanding of written and oral German
* Signed informed consent
* Scheduled for 24h blood pressure exam

Exclusion Criteria:

* Patients with unhealthy mental state
* Patients with an active implantable medical device (AIMD)
* Arteriopathy of the upper limbs with/without stenosis
* Severe congestive heart failure (LV-EF ≤25%)
* Sever aortic-valve stenosis mean gradient >40mmHg, valve area <1cm2)
* Congenital heart disease including aortic isthmus stenosis
* Untreated heart rhythm disorders, heart rate at rest > 120/bpm
* Severe untreated arterial hypertension (BPsyst > 180mmHg, BPdiast > 100mmHg)
* Atrial fibrillation
* Instable angina pectoris
* Malcompliance concerning medication intake
* Active alcohol or drug abuse
* Pregnancy or lactation (women of childbearing age will be asked to performed urinary pregnancy test before the screening phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the accuracy | Day 0 for 24 hours
  Continuous blood pressure measurement of the novel device will be compared to measurements assessed by a standard 24h blood pressure monitor at normal out of hospital conditions during night periods.

SECONDARY OUTCOMES:
Assessment of the acceptability | Day 1
  Acceptability of the novel blood pressure device in patients when used during 24 hours will be assessed by means of a questionnaire filled in by patients at day 1. The scale title is: Fragebogen. The minimum value is -1 and the maximum value is 10. The higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emrush Rexhaj, MD, Study Director — University Hospital Inselspital
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided